CLINICAL TRIAL: NCT06856174
Title: Menopausal Hormone Therapy for Women Living With HIV (HoT)
Brief Title: Menopausal HT for Women Living With HIV (HoT)
Acronym: HoT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Aging (NIA) (NIH); Exeltis (Industry); Xiromed LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5424; UM1AI068636 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-03-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HIV Infection; Menopause
MeSH Terms: conditions — HIV Infections | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Hormone Therapy (Active Comparator): PARTICIPANTS WITH INTACT UTERUS: Transdermal estradiol gel plus oral micronized progesterone daily for 12 weeks.
  PARTICIPANTS WITHOUT A UTERUS: Transdermal estradiol gel daily for 12 weeks.
  Interventions: Drug: Transdermal estradiol gel; Drug: Micronized Progesterone
- Arm B: Hormone Therapy Placebo (Placebo Comparator): PARTICIPANTS WITH INTACT UTERUS: Transdermal placebo gel plus oral encapsulated placebo pill daily for 12 weeks.
  PARTICIPANTS WITHOUT A UTERUS: Transdermal placebo gel alone daily for 12 weeks.
  Interventions: Drug: Placebo for estradiol gel; Drug: Placebo for micronized progesterone

INTERVENTIONS:
Drug: Transdermal estradiol gel — All participants: Estradiol gel 0.1%, 0.75 grams (corresponding to estradiol 0.75 mg) applied to the skin of the upper thigh once daily for 12 weeks.
  Arms: Arm A: Hormone Therapy
Drug: Micronized Progesterone — Participants with intact uterus: Encapsulated micronized progesterone 100 mg orally once daily for 12 weeks.
  Arms: Arm A: Hormone Therapy
Drug: Placebo for estradiol gel — All participants: Placebo for estradiol gel 0.1%, 0.75 grams applied to the skin of the upper thigh once daily for 12 weeks.
  Arms: Arm B: Hormone Therapy Placebo
Drug: Placebo for micronized progesterone — • Participants with intact uterus: Encapsulated placebo for micronized progesterone 100 mg orally once daily for 12 weeks.
  Arms: Arm B: Hormone Therapy Placebo

SUMMARY:
Women living with HIV have been shown to experience more frequent and severe hot flashes and night sweats (collectively known as vasomotor symptoms) as compared to women living without HIV. This correlates with disturbed sleep, increased depressive symptoms, increased anxiety, worse mental function, interference with activities of daily living including work, and worse overall quality of life.

Hormone therapy is considered to be the most effective therapy for hot flashes and night sweats and the most appropriate choice to prevent bone loss at the time of menopause for women without HIV. However, the usefulness of hormone therapy has not been specifically studied in women living with HIV.

This trial is being done to see if:

* There is evidence to support the use of hormone therapy (estradiol with or without progesterone) for the treatment of hot flashes and night sweats in women living with HIV
* Hormone therapy improves mental function, mood, sleep, quality of life, bone health, heart health, and inflammation in women living with HIV
* Hormone therapy is safe and tolerable for women living with HIV

ELIGIBILITY:
* Living with HIV
* Assigned female sex at birth
* Between the ages of 40 and 60 years
* In the late menopausal transition (perimenopause) or early postmenopause
* Experiencing hot flashes and/or night sweats
* Willing and able to complete a daily diary
* Does not have medical condition that would contraindicate hormone therapy
* Not taking medications to treat hot flashes
* Not taking medications that cannot be combined with hormone therapy
* Receiving antiretrovirals (HIV medication) for more than 1 year
* Not pregnant and willing and able to use at least non-hormonal birth control to prevent pregnancy
* Willing and able to provide informed consent after discussion with the research staff

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in vasomotor symptoms (VMS) frequency | From 5 weeks prior to randomization to Week 12
  Change in self-reported mean VMS frequency per day from 5-week observation phase prior to randomization to the one-week period prior to week 12 visit following.

SECONDARY OUTCOMES:
Change in vasomotor symptom (VMS) severity | From 5 weeks prior to randomization to week 12
  Change in self-reported mean severity of VMS from 5-week observation phase prior to randomization to the one-week period prior to week 12 visit following randomization; severity scale is ordinal: none (0), mild (1), moderate (2), severe (3).
Change in sleep | From randomization to week 12
  Change in total sleep scores from randomization visit to week 12 visit as measured by the Pittsburgh Sleep Quality Index (PSQI). Total sleep score determined by summing responses from seven assessments, where each assessment is scored from 0 (best) to 3 (worst). The minimum possible total sleep score is 0 (best) and the maximum possible score is 21 (worst). Higher total scores suggest more severe sleep problems. Change in total score calculated as Week 12 minus baseline. Negative change indicates better outcomes.
Change in insomnia | From randomization to week 12
  Change in total insomnia scores from randomization visit to week 12 visit as measured by the Insomnia Severity Index (ISI). Total insomnia score determined by summing responses from seven assessments, each rated on a Likert 5-point scale, where 0 indicates no problems and 4 indicates severe problems. The minimum possible total insomnia score is 0 (best) and the maximum possible score is 28 (worst). Higher total scores suggest more severe insomnia problems. Change in total score calculated as Week 12 minus baseline. Negative change indicates better outcomes.
Change in quality of life | From randomization to week 12
  Change in total health-related quality of life score, from randomization visit to week 12 visit as measured by Menopause specific Quality of life questionnaire (MenQOL). Total health-related quality of life score is determined by averaging responses from four domain-specific scores (vasomotor [3 items], physical [16 items], psychosocial [7 items], sexual functioning [3 items], each ranging from 1 (best) to 8 (worst)). Domain-specific scores represent the average score among the items in a domain. The score for each item, ranging from 1 (best) to 8 (worst), represents the sum of the presence of the symptom (1 for no, 2 for yes) and the severity, rated on a Likert 7-point scale (0, not bothered at all to 6, extremely bothered), The minimum possible quality of life score is 1 (best) and the maximum possible score is 8 (worst). Higher scores suggest more severe quality of life problems. Change in total score calculated as Week 12 minus baseline. Negative change indicates better outcomes.
Percentage of participants with adverse events associated with hormone therapy | From randomization to week 12
  Adverse events (AE) associated with study treatment with severity grade of 3 or higher as per DAIDS Toxicity grading scale.
Percentage of participants with occurrence of abnormal vaginal bleeding | From randomization to week 12
  Abnormal vaginal bleeding adverse event defined as any of the following: any report of heavy bleeding, 2 or more episodes of spotting or greater at intervals of < 21 days among participants in late menopausal transition, any occurrence after 6 weeks of hormone treatment among post-menopausal participants.
Percentage of participants with intolerance of hormone therapy | From randomization to week 12
  Intolerance of hormone therapy is defined as permanent discontinuation prior to the week 12 visit that was not required per protocol nor recommended due to safety considerations.
Change in neurocognitive test results | From randomization to week 12
  Change in neurocognition as measured by the neuropsychological (NP) battery from randomization visit to week 12 visit.
Change in depression symptoms | From randomization to week 12
  Change in depression symptoms score from randomization visit to week 12 visit as measured by Patient Health Questionnaire-9 (PHQ-9). Total depression score determined by summing responses from nine assessments, where each assessment is scored from 0 (not at all) to 3 (nearly every day). The minimum possible total sleep score is 0 (best) and the maximum possible score is 27 (worst). Higher total scores suggest more severe depression problems. Change in total score calculated as Week 12 minus baseline. Negative change indicates better outcomes.
Change in anxiety symptoms | From randomization to week 12
  Change in anxiety symptoms score from randomization visit to week 12 as measured by Generalized Anxiety Disorder 7-item (GAD-7). Total anxiety score determined by summing responses from seven Likert assessments, where each assessment is scored from 0 (best) to 3 (worst). The minimum possible total anxiety score is 0 (best) and the maximum possible score is 21 (worst). Higher total scores suggest more severe anxiety problems. Change in total score calculated as Week 12 minus baseline. Negative change indicates better outcomes.
Change in weight | From randomization to week 12
  Absolute and Percent change in total body weight from randomization visit to week 12 visit.
Change in body mass index (BMI) | From randomization to week 12
  Absolute change in BMI from randomization visit to week 12 visit
Change in waist circumference | From randomization to week 12
  Absolute change in minimum waist circumference from randomization visit to week 12 visit
Change in waist-to-hip ratio | From randomization to week 12
  Change in waist-to-hip circumference ratio between the randomization visit and the week 12 visit
Change in sexual function | From randomization to week 12
  Change in total sexual function score from randomization visit to week 12 visit as measured by the female sexual function index (FSFI). Total sexual function score is determined by summing six domain-specific scores (desire [2 items], arousal [4 items], lubrication [4 items], orgasm [3 items], satisfaction [3 items], and pain [3 items]), ranging from 0 (worst) to 6 (best). Domain-specific scores represent the sum of the scores for each item within a domain (ranging from 0 (worst) to 6 (best)), multiplied by a factor to adjust for relative weighting (0.6 for desire; 0.3 for arousal; 0.3 for lubrication; 0.4 for orgasm; 0.4 for satisfaction; and 0.4 for pain). The minimum possible sexual function score is 2 (worst) and the maximum possible score is 36 (best). Lower scores indicate worse sexual function. Change in total score calculated as Week 12 minus baseline. Positive change indicates better outcomes.
Percentage of participants with female sexual distress | Week 12 visit
  Female sexual distress defined as, at the week 12 visit, endorsing frequently or always to question regarding how often distressed or bothered about sex life in the past 4 weeks.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG).
  * For what types of analyses? To achieve aims in the proposal approved by the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG).
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections Group (ACTG) "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (ACTG) Data Use Agreement before receiving the data.